CLINICAL TRIAL: NCT05046795
Title: A Randomized, Double Blind, Placebo-Controlled, Parallel Group Study of Nebulized Revefenacin Inhalation Solution in Chinese Subjects With Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Revefenacin in Chinese Subjects With Moderate to Very Severe Chronic Obstructive Pulmonary Disease(COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Pharma UK Ltd. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REV-3001
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Results first posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: COPD
Keywords: Revefenacin; Long-acting muscarinic receptor antagonist(LAMA)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — revefenacin

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-blind, placebo-control, parallel group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Revefenacin inhalation solution 175 mcg QD. (Experimental): Revefenacin inhalation solution 175 mcg QD.
  Interventions: Drug: Revefenacin 175 mcg in 3 ML Inhalation Solution
- Placebo inhalation solution QD. (Placebo Comparator): Placebo inhalation solution QD.
  Interventions: Drug: Placebo inhalation solution QD

INTERVENTIONS:
Drug: Revefenacin 175 mcg in 3 ML Inhalation Solution — Revefenacin
  Arms: Revefenacin inhalation solution 175 mcg QD.
Drug: Placebo inhalation solution QD — Placebo
  Arms: Placebo inhalation solution QD.

SUMMARY:
This study is a phase III clinical study to assess the efficacy and safety of Revefenacin inhalation solution 175 mcg administered once daily via nebulization for 12 weeks compared to placebo in a population of Chinese subjects with moderate to very severe COPD.

DETAILED DESCRIPTION:
This will be a multi-center, randomized, double blind, placebo-controlled, parallel group study, randomizing approximately 320 male or female moderate-very severe COPD subjects. Subjects will receive study drug for 12 weeks. Treatments to be received during the study will include one of the following, administered using a centrally-provided, standard jet nebulizer and compressor via a mouthpiece: A. Revefenacin inhalation solution 175 mcg Quaque die (QD). B. Placebo inhalation solution QD. Subjects will have approximately 6 clinic visits (encompassing a screening period of up to 30 days and a treatment period of 12 weeks), and a follow-up telephone call 1-2 weeks after the End of Treatment (EoT) visit.

ELIGIBILITY:
Inclusion Criteria:

* Key inclusion criteria include:

  * Males and females of Chinese ethnicity, at least 40 years of age. Females may be of either childbearing or non-childbearing potential. All females of childbearing potential must be using an acceptable, highly effective method of contraception and have a negative pregnancy test at screening.
  * A clinical diagnosis for at least 6 months prior to screening of COPD according to Global Initiative for Chronic Obstructive Lung Disease(GOLD) guidelines.
  * Subject is capable of performing reproducible spirometry maneuvers as described by current American Thoracic Society/European Respiratory Society (ATS/ERS) Guidelines and has a post-ipratropium (500 mcg nebulized) Forced Expiratory Volume in

    1 second(FEV1)/Forced Vital Capacity(FVC) ratio <0.7 at Visit 2.
  * Subject has moderate to very severe COPD with a post-ipratropium (500 mcg nebulized) FEV1 less than 80% of predicted normal (using the Global Lung Function Initiative reference range; ) and an absolute FEV1 >700 mL at Visit 2
  * Current smoker or ex-smoker, with a history of at least 10 pack-years of tobacco smoking. Ex-smokers must have stopped smoking >6 months prior to Visit 1.

Exclusion Criteria:

* Key exclusion criteria include:

  * Previously dosed with Revefenacin.
  * Current diagnosis of asthma.
  * Alpha-1 anti-trypsin deficiency.
  * Other chronic or active respiratory disorder (e.g., clinically significant [as determined by the Investigator] bronchiectasis, pulmonary fibrosis, sarcoidosis, pneumoconiosis, active tuberculosis).
  * Symptoms of, or treatment for an Acute Exacerbation of COPD(AECOPD) requiring antibiotics and/or oral/systemic corticosteroids or in-patient hospitalization during the 28 days preceding screening or during the screening period between Visit 1 and Visit 3.
  * Pneumonia requiring hospitalization within 28 days prior to screening or during the screening period between Visit 1 and Visit 3.
  * Lower respiratory tract infection requiring treatment with antibiotics during the 28 days preceding screening or during the screening period between Visit 1 and Visit 3.
  * History or presence of pulmonary hypertension, respiratory failure, cor pulmonale or right ventricular failure which may impact the safety of the subject in the clinical judgement of the Investigator.
  * History of pulmonary lobectomy, lung volume reduction surgery, or lung transplantation.
  * Use of supplemental oxygen therapy for more than 15 hours per day (includes night-time use).
  * Subjects with hepatic impairment.
  * Subject suffers from any medical condition that would preclude the use of inhaled anticholinergics, including narrow-angle glaucoma, symptomatic benign prostatic hyperplasia, bladder neck obstruction, or urinary retention.
  * Subjects who are unable to stop any of the following medications, and refrain from their use throughout the study until the final dose of study drug:

    * Short-acting β2 agonists (except study-supplied salbutamol).
    * Short-acting anticholinergic agents (except those used for reversibility testing).
    * Long-acting anticholinergics (except study supplied medication).
    * Combination β2 agonists/anticholinergic agents.
    * Combination β2 agonists/inhaled corticosteroids/anticholinergic agents.
    * Phosphodiesterase 4 inhibitors.
    * Theophyllines.
    * Leukotriene inhibitors.
    * Orally inhaled nedocromil or cromolyn sodium.
    * Oral or parenteral corticosteroids.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dik WH Ng, PhD, Study Director — Mylan Pharmaceuticals Inc
Locations (35):
- China (35):
  - Anhui Medical University - Hefei First People's Hospital, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - The Third Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The Second Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Gunagdong
  - Hainan General Hospital, Haikou, Hainan
  - The First Hospital of Changsha, Changsha, Hunan
  - Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia
  - The First Affiliated Hospital of Baotou Medical College - Respiration, Baotou, Inner Mongolia
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - Affiliated Hospital of Inner Mongolia Medical College, Hohhot, Inner Mongolia
  - Jiangsu Jiangyin People's Hospital, Jiangyin, Jiangsu
  - Zhongda Hospital, Southeast University - Pulmonology, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Yangzhou First People's Hospital, Yangzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Nanchang University - The Second Affiliated Hospital, Nanchang, Jiangxi
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Yanbian university hospital, Yanji, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area People's Hospital, Shanghai, Shanghai Municipality
  - Sichuan University - West China Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital - Respiration, Tianjin, Tianjin Municipality
  - The First Center hospital of Tianjin, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University - Hospital, Ürümqi, Xinjiang
  - Dongyang People's Hospital, Dongyang, Zhejiang
  - Xinhua Hostipal of Zhejiang Province, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 258 subjects were randomized, of which 257 received randomized study treatment. The one subject who was not treated was randomized in error
Groups:
- Revefenacin Inhalation Solution 175 mcg QD.: Revefenacin inhalation solution 175 mcg in 3 mL administered once daily by nebulizer for 12 weeks
- Placebo Inhalation Solution QD.: Placebo inhalation solution in 3 mL administered once daily by nebulizer for 12 weeks
Period: Overall Study
Arm/Group | Revefenacin Inhalation Solution 175 mcg QD. | Placebo Inhalation Solution QD.
Started (Subjects who received at least one dose of study treatment) | 129 | 128
Completed | 107 | 99
Not Completed | 22 | 29
Not completed — Adverse Event | 13 | 15
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Death | 1 | 0
Not completed — Public health emergency (COVID-19) restrictions | 2 | 3

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS), which consisted of all randomized subjects who received at least one dose of study drug and had at least one recorded post-baseline efficacy assessment. Subjects in this set were analyzed and summarized according to their assigned treatment and strata at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Revefenacin Inhalation Solution 175 mcg QD. | Placebo Inhalation Solution QD. | Total
Number analyzed (Participants) | 129 | 128 | 257
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.6 (6.18) | 67.7 (6.80) | 67.6 (6.48)
Age, Customized [Count of Participants; unit: Participants]
  Age group: <65 years | 36 | 37 | 73
  Age group: >=65 years | 93 | 91 | 184
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 122 | 122 | 244
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian - Chinese | 129 | 128 | 257
  Race: Asian - Not Chinese | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 129 | 128 | 257
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.92 (3.559) | 23.44 (3.106) | 23.18 (3.345)
Concomitant inhaled corticosteroid use [Count of Participants; unit: Participants]
  Yes | 85 | 88 | 173
  No | 44 | 40 | 84
Concomitant long acting beta agonist use [Count of Participants; unit: Participants]
  Yes | 87 | 87 | 174
  No | 42 | 41 | 83
Reversibility to ipratropium [Count of Participants; unit: Participants] — Bronchodilator reversibility was performed at screening with ipratropium 500 mcg solution for inhalation administered by jet nebulizer, after withholding short-acting bronchodilators for at least 6 hours. Spirometry was performed pre-dose and 45 minutes after dosing with ipratropium. Reversibility to ipratropium was defined as a post-bronchodilator increase of ≥12% and at least a 200 mL increase in FEV1.
  Participants
    Yes | 59 | 57 | 116
    No | 70 | 71 | 141

OUTCOME MEASURES:

1. Primary Outcome: Trough FEV1 on Day 85
Description: Change from Baseline (Day 1, pre-dose) trough FEV1 on Day 85
Time Frame: Baseline and Day 85
Population: The Analysis Population was all subjects in the Full Analysis Set who had evaluable data for the respective endpoint. Missing data was not imputed.
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Revefenacin Inhalation Solution 175 mcg QD. | Placebo Inhalation Solution QD.
Number analyzed (Participants) | 105 | 99
mL | 55.12 (23.974) | -95.78 (24.504)
Statistical Analysis 1: Comparison: Revefenacin Inhalation Solution 175 mcg QD. vs Placebo Inhalation Solution QD; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 150.91, 95% CI 2-sided [104.145 to 197.671], Standard Error of Mean 23.727

2. Primary Outcome: Trough FEV1 on Day 85 - Sensitivity Analysis With Missing Data Imputed
Description: Sensitivity analysis results of change from baseline in trough FEV1 (mL) on Day 85 with missing data imputed by last observation carried forward
Time Frame: Baseline, Day 29, Day 57 and Day 85
Population: Full analysis set (missing data for Day 85 was imputed from Day 29 or Day 57 data by Last Observation Carried Forward)
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Revefenacin Inhalation Solution 175 mcg QD. | Placebo Inhalation Solution QD.
Number analyzed (Participants) | 129 | 128
mL | 52.05 (27.036) | -92.30 (27.502)
Statistical Analysis 1: Comparison: Revefenacin Inhalation Solution 175 mcg QD. vs Placebo Inhalation Solution QD; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 144.35, 95% CI 2-sided [102.610 to 186.088], Standard Error of Mean 21.192

3. Secondary Outcome: Trough FVC on Day 85
Description: Change from baseline (Day 1, pre-dose) trough Forced Vital Capacity (FVC) on Day 85
Time Frame: Baseline and Day 85
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Revefenacin Inhalation Solution 175 mcg QD. | Placebo Inhalation Solution QD.
Number analyzed (Participants) | 105 | 99
mL | 97.92 (41.833) | -189.83 (42.801)
Statistical Analysis 1: Comparison: Revefenacin Inhalation Solution 175 mcg QD. vs Placebo Inhalation Solution QD; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 287.75, 95% CI 2-sided [211.933 to 363.570], Standard Error of Mean 38.473

4. Secondary Outcome: Change From Baseline in Peak FEV1 (0-2h) on Day 1
Description: Baseline FEV1 was defined as the average of the -45 and -15 minute measurements prior to dosing of study drug on Day 1. Peak FEV1 (0-2h) was defined as the highest post dose FEV1 value within 2 hours after the dosing.
Time Frame: Day 1, from 45 minutes before dosing to 2 hours after dosing
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Revefenacin Inhalation Solution 175 mcg QD. | Placebo Inhalation Solution QD.
Number analyzed (Participants) | 129 | 128
mL | 234.2 (21.55) | 128.4 (21.92)
Statistical Analysis 1: Comparison: Revefenacin Inhalation Solution 175 mcg QD. vs Placebo Inhalation Solution QD; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Net) = 105.9, 95% CI 2-sided [72.60 to 139.12], Standard Error of Mean 16.89

5. Secondary Outcome: Change From Baseline in Peak FEV1 (0-2h) on Day 85
Description: as for outcome 4
Time Frame: Day 1 (baseline) and Day 85, from 45 minutes before dosing to 2 hours after dosing
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Revefenacin Inhalation Solution 175 mcg QD. | Placebo Inhalation Solution QD.
Number analyzed (Participants) | 103 | 97
mL | 199.0 (32.72) | 44.2 (33.62)
Statistical Analysis 1: Comparison: Revefenacin Inhalation Solution 175 mcg QD. vs Placebo Inhalation Solution QD; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Net) = 154.8, 95% CI 2-sided [98.86 to 210.78], Standard Error of Mean 28.37

6. Secondary Outcome: Change From Baseline in SGRQ Total Score on Day 85
Description: Change from Baseline in the St George's Respiratory Questionnaire (SGRQ) Total Score on Day 85.
  Scores range from 0 to 100, with higher scores indicating more health limitations. A reduction of 4 or more points is considered to be a clinically meaningful improvement
Time Frame: Day 1 (baseline) and Day 85
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Revefenacin Inhalation Solution 175 mcg QD. | Placebo Inhalation Solution QD.
Number analyzed (Participants) | 110 | 112
Score on a scale | -4.8 (2.17) | 0.2 (2.20)
Statistical Analysis 1: Comparison: Revefenacin Inhalation Solution 175 mcg QD. vs Placebo Inhalation Solution QD; Test type: Superiority; p = 0.0064, ANCOVA; Mean Difference (Net) = -4.9, 95% CI 2-sided [-8.49 to -1.40], Standard Error of Mean 1.80

7. Secondary Outcome: Number (%) of SGRQ Responders on Day 85
Description: Number of subjects with a decrease from baseline of ≥4 units in SGRQ total score (which was defined as a responder) on Day 85
Time Frame: Day 85
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Revefenacin Inhalation Solution 175 mcg QD. | Placebo Inhalation Solution QD.
Number analyzed (Participants) | 110 | 112
Participants | 58 | 45
Statistical Analysis 1: Comparison: Revefenacin Inhalation Solution 175 mcg QD. vs Placebo Inhalation Solution QD; Test type: Superiority; p = 0.0144, Regression, Logistic; Odds Ratio (OR) = 2.1, 95% CI 2-sided [1.16 to 3.84]

ADVERSE EVENTS:
Time Frame: 12 week treatment period and for up to 30 days after the last dose of study drug
Arm/Group | Revefenacin Inhalation Solution 175 mcg QD. | Placebo Inhalation Solution QD.
All-Cause Mortality (participants affected / at risk) | 1/129 | 0/128
Serious Adverse Events (participants affected / at risk) | 14/129 | 11/128
Other Adverse Events (participants affected / at risk) | 58/129 | 60/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revefenacin Inhalation Solution 175 mcg QD. (N=129) | Placebo Inhalation Solution QD. (N=128)
COPD (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
HIV infection (Infections and infestations) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Cor pulmonale chronic (Cardiac disorders) | 1 (1) | 0 (0)
Postauricular fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Prostatic disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revefenacin Inhalation Solution 175 mcg QD. (N=129) | Placebo Inhalation Solution QD. (N=128)
COVID-19 (Infections and infestations) | 12 (12) | 8 (8)
Pneumonia (Infections and infestations) | 5 (5) | 3 (3)
Coronavirus infection (Infections and infestations) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 11 (13)
Asymptomatic bacteriuria (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
COPD (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 15 (15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chest discomfort (General disorders) | 8 (9) | 5 (5)
Pyrexia (General disorders) | 4 (4) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Asthenopia (Eye disorders) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Renal cyst (Renal and urinary disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 3 (3)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication by an Institution/Investigator of the study results shall not be made before the first multi-center publication by the Sponsor.

Thereafter, before submission for publication or presentation, the Investigator shall allow the Sponsor at least 60 days to review any manuscript and at least 30 days to review any poster presentation, abstract or other written or oral material. The Sponsor may request in writing that any publication or presentation be withheld for a further 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT05046795/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT05046795/SAP_001.pdf